CLINICAL TRIAL: NCT01585857
Title: A Phase I, Prospective, Bi-centric,Single -Arm, Open-label, Dose-escalating Clinical Trial to Evaluate the Safety of a Single Injection of Autologous Adipose Derived Mesenchymal Stromal Cells in the Treatment of Severe Osteoarthritis of the Knee Joint
Brief Title: ADIPOA - Clinical Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8606
Record Dates: First submitted 2012-03-19; First posted 2012-04-26 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): 2 x 10E6 ASC intra-articular injection (5 ml)
  Interventions: Biological: Autologous adipose derived stem cells administrated for intra-articular use
- Group 2 (Experimental): 10 x 10E6 ASC intra-articular injection (5 ml)
  Interventions: Biological: Autologous adipose derived stem cells administrated for intra-articular use
- Group 3 (Experimental): 50 x 10E6 ASC intra-articular injection (5 ml)
  Interventions: Biological: Autologous adipose derived stem cells administrated for intra-articular use

INTERVENTIONS:
Biological: Autologous adipose derived stem cells administrated for intra-articular use — Each patient will receive one single administration of the cells and will be followed for 3 months. Each patients will be follow-up during one year with routinely examinations for safety issues.
  Arms: Group 2; Group 3
Biological: Autologous adipose derived stem cells administrated for intra-articular use — Each patient will receive one single administration of the cells and will be followed for 3 months. Each patients will be follow-up during one year with routinely examinations for safety issues. The first patient will be followed during 12 weeks before inclusion of the second patient.
  Arms: Group 1

SUMMARY:
Primary:

To study the safety of a single injection of autologous adipose derived mesenchymal stromal cells (ASCs) on patients with moderate or severe osteoarthritis of the knee (OA).

Secondary:

To study the efficacy of a single injection of autologous adipose derived mesenchymal stromal cells on patients with moderate or severe osteoarthritis of the knee (OA).

ELIGIBILITY:
Inclusion Criteria:

* OA diagnosis should fulfil the criteria of the American College of Rheumatology (ACR) with moderate or severe medial and/ or external femorotibial knee osteoarthritis (OA) (stage 3 or 4) and indication total knee arthroplasty.

Exclusion Criteria:

* Any disease or medication affecting the bone or cartilage metabolism, including corticoids.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Recording of Serious Adverse Events | during 365 days following injection
  Adverse events will be described with respect to seriousness, intensity, relationship to treatment, action taken and outcome of the adverse event.

SECONDARY OUTCOMES:
Functional status of the knee | during 365 days following injection
  Efficacy will be assessed by measuring:
  * WOMAC (Western Ontario and McMaster Universities osteoarthritis index),
  * Short Arthritis assessment Scale (SAS),
  * range of motion of the target knee joint,
  * imaging through MRI evaluation, dGEMRIC and T1rho MRI.
Evaluation of Quality of life | during 365 days following injection
  Quality of life will be assessed by measuring:
  * pain-specific assessment
  * global patient assessment (visual analog scale, Short-Form 8)
  * decrease in rescue paracetamol medication.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jorgensen, MD, Principal Investigator — University Hospital, Montpellier
Locations (2):
- UH Montpellier, Montpellier, France
- Orthopädische Klinik, Würzburg, Germany

REFERENCES:
- [Derived] Pers YM, Rackwitz L, Ferreira R, Pullig O, Delfour C, Barry F, Sensebe L, Casteilla L, Fleury S, Bourin P, Noel D, Canovas F, Cyteval C, Lisignoli G, Schrauth J, Haddad D, Domergue S, Noeth U, Jorgensen C; ADIPOA Consortium. Adipose Mesenchymal Stromal Cell-Based Therapy for Severe Osteoarthritis of the Knee: A Phase I Dose-Escalation Trial. Stem Cells Transl Med. 2016 Jul;5(7):847-56. doi: 10.5966/sctm.2015-0245. Epub 2016 May 23. PMID 27217345